CLINICAL TRIAL: NCT05831696
Title: Metabolic Cost of Walking With Passive vs. Powered Prosthetic Knees Among Persons With Limb Loss
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Collaborators: Össur Iceland ehf (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 5220320
Record Dates: First submitted 2023-02-27; First posted 2023-04-26 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Transfemoral Amputation
Keywords: Power Knee; Amputation; Metabolic Costs; Heart Rate

STUDY DESIGN:
Intervention Model Description: Participants will be their own control
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Powered Microprocessor-controlled Knee (PMPK) (Experimental): the "Power Knee" is a commercially available PMPK.
  Interventions: Other: Powered Microprocessor-controlled Knee (PMPK)

INTERVENTIONS:
Other: Powered Microprocessor-controlled Knee (PMPK) — A microprocessor-controlled Knee with standardized commercial prosthetic foot
  Other Names: Power Knee

SUMMARY:
The purpose of this industry-initiated research study is to test that a powered microprocessor controlled knee improves metabolic function during walking in level and sloped conditions as compared to the subject's physician prescribed prosthesis.

DETAILED DESCRIPTION:
The Procedures include:

Initial Visit:

1. Informed consent
2. HIPAA authorization
3. Determine/verify ambulation potential
4. Take and record body measurements (height, weight, circumferences)
5. Activities-Specific Balance Confidence (ABC) scale
6. L.A.S.A.R. Posture alignment assessment with RxPx

Second Visit

1. Fit with heartrate monitor and metabolic analyzer mask
2. Treadmill Test (level-ground) with RxPx
3. Rest
4. Treadmill Test (incline) with RxPx
5. Fit subject with PMPK
6. L.A.S.A.R. Posture alignment assessment with PMPK
7. Subject uses PMPK for one week as their primary prosthesis

Third Visit (1 week later)

1. Fit with heartrate monitor and metabolic analyzer mask
2. Treadmill Test (level-ground) with PMPK
3. Rest
4. Treadmill Test (incline) with PMPK
5. Activities-Specific Balance Confidence (ABC) scale
6. Return PMPK and refit of RxPx
7. Verify alignment with L.A.S.A.R. Posture alignment
8. Check that all fasteners are secure

ELIGIBILITY:
Inclusion Criteria:

* Males and Females with unilateral knee disarticulation or transfemoral (KD/TF) amputation.
* a body mass greater than 49Kg and less than 117Kg
* 18-75 years of age
* Have an ambulation potential of K3 or K4
* Use a prosthesis daily for walking or sports activities
* No less than six months of experience with a prosthesis
* No socket issues or changes in the last six weeks
* No residual limb pain affecting functional ability.

Exclusion Criteria:

* Cannot walk at different speeds (MCFL K0-K2)
* Limb-loss below the knee or through the hip
* More than one amputation.
* Uses an assistive device for walking
* Uncontrolled edema in leg compartments
* Compromised skin of the residual limb or contralateral foot
* Are 180 days or less post-amputation
* Pregnant (self-reported)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-02-27 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
VO2 uptake - level ground | Change between Baseline Visit (study enrollment) and Visit 2 (3 weeks post-study enrollment)
  VO2 uptake during ambulation on a treadmill - level ground
VO2 uptake - incline | Visit 2 (3 weeks post-study enrollment)
  VO2 uptake during ambulation on a treadmill - 5 degree incline

SECONDARY OUTCOMES:
Balance confidence | At Baseline Visit (study enrollment)
  Activities based balance confidence survey (0-100%) higher score means more balance confidence
Exertion | Change between Visit 2 (3 weeks post-study enrollment) and Visit 3 (4 weeks post-study enrollment)
  Borg Exertion Scale (0-10) with 10 being maximum exertion

CONTACTS AND LOCATIONS:
Overall Officials: Michael Davidson, Ph.D., Principal Investigator — Loma Linda University Health
Locations (1):
- Loma Linda University, Loma Linda, California, United States